CLINICAL TRIAL: NCT06251154
Title: A Clinical Comparison of Two Soft Contact Lenses (Iteration Under Umbrella Protocol C19-678)
Brief Title: Clinical Comparison of Two Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-154
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (Experimental): All participants wore Lens 1 for 15 minutes (Period 1)
  Interventions: Device: Lens 1
- Lens 2 (Experimental): All participants wore Lens 2 for 15 minutes (Period 2)
  Interventions: Device: Lens 2

INTERVENTIONS:
Device: Lens 1 — Daily disposable silicone hydrogel contact lens (diameter=14.0mm) for 15 minutes
  Arms: Lens 1
Device: Lens 2 — Daily disposable silicone hydrogel contact lens (diameter=14.1mm) for 15 minutes
  Arms: Lens 2

SUMMARY:
This study was designed to gather short-term clinical performance data for 2 soft contact lenses.

DETAILED DESCRIPTION:
The purpose of this participant-masked, non-randomized, crossover controlled, non-dispensing, study was to compare the short-term performance of 2 daily disposable contact lenses after 15 minutes of daily wear each. The lenses were identical in all aspects except for diameter. Participants attended for 1 visit only which lasted for approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They were of legal age (18) and capacity to volunteer.
  2. They understood their rights as a research subject and were willing and able to sign a Statement of Informed Consent.
  3. They were willing and able to follow the protocol.
  4. They were wearing soft contact lenses, or had done so within the past two years.
  5. They were able to be fitted with the study lenses within the power range available.

Exclusion Criteria:

* Subjects will not be eligible if:

  1. They had an ocular disorder which would normally contra-indicate contact lens wear.
  2. They had a systemic disorder which would normally contra-indicate contact lens wear.
  3. They were using any topical medication such as eye drops or ointment.
  4. They were aphakic.
  5. They had had corneal refractive surgery.
  6. They had any corneal distortion resulting from previous hard or rigid lens wear or had keratoconus.
  7. They were pregnant or lactating.
  8. They had an eye or health condition including an immunosuppressive or infectious disease which could, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
  9. They had taken part in any contact lens or care system clinical research within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, PhD MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Period 1: Lens 1, 15 Minutes
Arm/Group | Lens 1 | Lens 2
Started | 50 | 0 (All participants received Lens 1 in Period 1.)
Completed | 50 | 0
Not Completed | 0 | 0
Period: Period 2: Lens 2, 15 Minutes
Arm/Group | Lens 1 | Lens 2
Started | 0 (All participants received Lens 2 in Period 2.) | 50
Completed | 0 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who participated in the clinical trial.
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data is presented as stratified by the sex of the participant
  years | 37.9 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Score
Description: Subjective overall score was assessed using 0-100 visual analogue scale, where 0=Extremely poor, unmanageable, cannot use lenses and 100=Excellent, highly impressed with these lenses overall
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens 1: All participants that received Lens 1
- Lens 2: All participants that received Lens 2
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 50 | 50
score on a scale | 80.2 (16.7) | 88.2 (11.0)

2. Secondary Outcome: Subjective Comfort
Description: Subjective comfort score was assessed using 0-100 visual analogue scale, where 0=Extremely uncomfortable, causes pain, cannot be tolerated and 100=Excellent, cannot be felt
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 50 | 50
score on a scale | 81.1 (20.1) | 90.4 (9.6)

3. Secondary Outcome: Subjective Vision
Description: Subjective vision score was assessed using a 0-100 visual analogue scale, where 0=Extremely poor, intolerable, lens cannot be worn and 100=Excellent, unaware of any visual loss
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 50 | 50
score on a scale | 81.9 (16.1) | 87.2 (12.6)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 hours
Arm/Group | Lens 1 | Lens 2
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT06251154/Prot_SAP_000.pdf